CLINICAL TRIAL: NCT00688545
Title: SINCERE™: Safety in Idiopathic Arthritis: NSAIDs and Celebrex Evaluation Registry A Prospective Observational Registry Of Patients With Juvenile Idiopathic Arthritis (JIA) Treated With NSAIDs
Brief Title: Naturalistic Safety Registry Of Celecoxib (CELEBREX(R)) And NSAIDs In Juvenile Idiopathic Arthritis
Acronym: SINCERE
Status: Terminated | Type: Observational
Why Stopped: See termination reason in detailed description.
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Other Study IDs: A3191344
Record Dates: First submitted 2008-05-29; First posted 2008-06-03 (Estimated); Results first posted 2013-07-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Arthritis, Juvenile Rheumatoid
Keywords: Celecoxib; COX-2; NSAIDs; observational study; noninterventional study; cohort study; registry; epidemiologic study; pediatrics; rheumatology; phase iv study
MeSH Terms: conditions — Arthritis, Juvenile | interventions — Celecoxib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Celecoxib: Patients treated with celecoxib as per treating physician's judgement
  Interventions: Drug: Celecoxib
- nsNSAIDs (nonselective nonsteroidal anti-inflammatory drugs): Patients treated with nsNSAIDs as per treating physician's judgement
  Interventions: Drug: nsNSAIDs

INTERVENTIONS:
Drug: Celecoxib — Non-interventional: Treatment assignment as per treating physician's judgement
  Groups: Celecoxib
Drug: nsNSAIDs — Non-interventional: Treatment assignment as per treating physician's judgement
  Groups: nsNSAIDs (nonselective nonsteroidal anti-inflammatory drugs)

SUMMARY:
This multi-center observational Registry will collect long-term safety data on patients treated with celecoxib or non-selective nonsteroidal anti-inflammatory drugs (nsNSAIDs) as used in clinical practice for the treatment of Juvenile Idiopathic Arthritis (JIA).

DETAILED DESCRIPTION:
None Study has been terminated early (LSLV = 09Jan2012) due to release of the postmarketing commitment by the US FDA. The study was stopped for futility/change in treatment paradigm that minimizes chronic NSAID use and not for safety concerns.

ELIGIBILITY:
Inclusion Criteria:

* Age at least 2 years but less than 18 years; JIA of any of the following subtypes: oligoarthritis, polyarthritis, or stable systemic disease;
* new treatment (started not more than 6 months prior) with one NSAID (celecoxib or nsNSAID).

Exclusion Criteria:

* Patients with the following JIA subtypes: active systemic disease, psoriatic Arthritis, enthesitis-related Arthritis, or undifferentiated arthritis;
* Patients with Reiter's syndrome; patients unlikely to complete 2 years of follow up;
* Patients who need to use multiple NSAIDs at the same time.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Juvenile Idiopathic Arthritis (JIA) subtypes that correspond to the former Juvenile Rheumatoid Arthritis (JRA) classification system who are treated by a participating pediatric rheumatologist and treated with either celecoxib or an nsNSAID; celecoxib or nsNSAID must be new treatment or recent initiation (within last 6 months).
Sampling Method: Non-Probability Sample
Enrollment: 275 (Actual)
Dates: Start 2009-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (26):
- United States (26):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Little Rock, Arkansas
  - Pfizer Investigational Site, Washington D.C., District of Columbia
  - Pfizer Investigational Site, Arlington Heights, Illinois
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Glenview, Illinois
  - Pfizer Investigational Site, New Lenox, Illinois
  - Pfizer Investigational Site, Westchester, Illinois
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Hackensack, New Jersey
  - Pfizer Investigational Site, Livingston, New Jersey
  - Pfizer Investigational Site, Brooklyn, New York
  - Pfizer Investigational Site, Commack, New York
  - Pfizer Investigational Site, Great Neck, New York
  - Pfizer Investigational Site, New Hyde Park, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Durham, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Liberty Township, Ohio
  - Pfizer Investigational Site, Mayfield Heights, Ohio
  - Pfizer Investigational Site, Strongsville, Ohio
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Charleston, South Carolina
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, Austin, Texas

REFERENCES:
- [Derived] Sobel RE, Lovell DJ, Brunner HI, Weiss JE, Morris PW, Gottlieb BS, Chalom EC, Jung LK, Onel KB, Petiniot L, Goldsmith DP, Nanda K, Shishov M, Abramsky S, Young JP, Giannini EH; Pediatric Rheumatology Collaborative Study Group. Safety of celecoxib and nonselective nonsteroidal anti-inflammatory drugs in juvenile idiopathic arthritis: results of the Phase 4 registry. Pediatr Rheumatol Online J. 2014 Jul 16;12:29. doi: 10.1186/1546-0096-12-29. eCollection 2014. PMID 25057265
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3191344&StudyName=Naturalistic%20Safety%20Registry%20Of%20Celecoxib%20%28CELEBREX%28R%29%29%20And%20NSAIDs%20In%20Juvenile%20Idiopathic%20Arthritis

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 275 people consented to participate in this study. One person should not have been enrolled and instead should have been a screen failure. This person did not receive any study drug.
Groups:
- Celecoxib: Participants who were prescribed celecoxib at baseline per treating physician's judgment. Participants could switch to nonselective non-steroidal anti-inflammatory drugs (nsNSAIDs) at any time during the study. The use and dosage recommendations for celecoxib took place on the basis of the approved Product Label and were adjusted solely according to medical and therapeutic necessity.
- nsNSAIDs: Participants who were prescribed nsNSAIDs at baseline per treating physician's judgment. Any nsNSAID could be used at the discretion of the investigator, provided that the medicine was not contraindicated for the participant as per the current United States product information for that nsNSAID. Participants could switch to other nsNSAIDs or celecoxib at any time during the study. The use and dosage recommendations for study drug took place on the basis of the approved Product Label and were adjusted solely according to medical and therapeutic necessity.
Period: Overall Study
Arm/Group | Celecoxib | nsNSAIDs
Started | 55 | 219
Switched Treatment at Least Once | 6 | 13
Completed | 50 | 204
Not Completed | 5 | 15
Not completed — Lost to Follow-up | 1 | 4
Not completed — Insurance/cost of drug | 0 | 1
Not completed — Withdrawal by Subject | 2 | 3
Not completed — Unspecified, unrelated to AE/Toxicity | 2 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Celecoxib | nsNSAIDs | Total
Number analyzed (Participants) | 55 | 219 | 274
Age, Customized [Number; unit: Participants]
  2-5 years | 8 | 77 | 85
  6-9 years | 17 | 52 | 69
  10-12 years | 15 | 44 | 59
  13-15 years | 7 | 35 | 42
  16-18 years | 8 | 11 | 19
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 165 | 212
  Male | 8 | 54 | 62
Juvenile Idiopathic Arthritis (JIA) [Number; unit: Participants] — Number of participants with JIA by subtype: systemic persistent oligoarticular, extended oligoarticular, polyarticular rheumatoid factor negative (Poly RF-) and positive (Poly RF+).
  Participants
    Systemic | 0 | 3 | 3
    Persistent Oligoarticular | 27 | 119 | 146
    Extended Oligoarticular | 2 | 12 | 14
    Poly RF- | 23 | 70 | 93
    Poly RF+ | 3 | 14 | 17
    Missing | 0 | 1 | 1
Gastrointestinal Symptom Scale for Kids (GISSK) - Type of stomach problems [Number; unit: Participants] — Participant or caregiver reported severity of participant's stomach problems during the last week using visual analogue scale (VAS), scores ranged from 0 (no trouble at all) to 100 (severe stomach problems). Also identified types of participant's stomach problems, if any, during the last week by selecting one or more check boxes.
  Participants
    Heartburn | 9 | 21 | 30
    Upper stomach pain | 8 | 18 | 26
    Lower stomach pain | 16 | 34 | 50
    Nausea | 14 | 32 | 46
    Diarrhea | 5 | 18 | 23
    Constipation | 5 | 16 | 21
    Vomiting | 2 | 8 | 10
    Poor appetite | 7 | 13 | 20
    No problems | 23 | 132 | 155
    Missing | 1 | 3 | 4
JIA medications [Number; unit: Participants] — JIA medications by class: GI protective agents (eg, proton-pump inhibitors), other GI, DMARDs, biologics, antihypertensives, NSAIDs (Celecoxib, Diclofenac, Ibuprofen, Meloxicam, Naproxen, other), corticosteroids (oral, intravenous [IV], intra-articular, other forms), analgesics (eg, Acetaminophen). Participants could receive more than 1 medication.
  Participants
    Gastrointestinal (GI) protective agents | 18 | 48 | 66
    Other GI | 4 | 4 | 8
    Disease-modifying antirheumatic drugs (DMARDs) | 21 | 83 | 104
    Biologics | 8 | 28 | 36
    Antihypertensives | 1 | 4 | 5
    NSAIDs (Celecoxib) | 8 | 0 | 8
    NSAIDs (Diclofenac) | 0 | 0 | 0
    NSAIDs (Ibuprofen) | 2 | 7 | 9
    NSAIDs (Meloxicam) | 0 | 6 | 6
    NSAIDs (Naproxen) | 0 | 16 | 16
    NSAIDs (Other) | 0 | 5 | 5
    Corticosteroids (Oral, IV, Intra-Articular) | 5 | 19 | 24
    Corticosteroids (Other) | 2 | 3 | 5
    Analgesics (Acetaminophen, Opioids, Other) | 9 | 18 | 27
Number of participants with abnormal physical exam results [Number; unit: Participants] — Abnormal findings in physical examination as determined by physician
  Participants | 17 | 63 | 80
Physician Global Assessment (PGA) of Disease Activity [Mean (Standard Deviation); unit: Units on a scale] — PGA measured on a scale from 0 (not active) to 10 (very active) where higher scores indicated more disease activity.
  Units on a scale | 2.6 (2.36) | 2.9 (2.19) | 2.8 (2.22)
Participant or caregiver's assessment of participant's overall well-being [Mean (Standard Deviation); unit: Units on a scale] — Overall well being measured on a scale from 0 (very well) to 10 (very poor).
  Units on a scale | 3.2 (2.58) | 2.8 (2.50) | 2.9 (2.52)
Child Health Questionnaire (CHAQ) - global evaluation [Mean (Standard Deviation); unit: Units on a scale] — CHAQ: validated parent or legal guardian assessed instrument of child's activities of daily living, pain, and global assessment. Global evaluation rated on a visual analog scale (VAS) from 0 (very well) to 100 (very poor) where higher scores indicated a worse evaluation.
  Units on a scale | 29.11 (29.34) | 20.15 (21.58) | 21.96 (23.56)
CHAQ - pain [Mean (Standard Deviation); unit: Units on a scale] — CHAQ: validated parent or legal guardian assessed instrument of child's activities of daily living, pain, and global assessment. Pain rated on a VAS from 0 (no pain) to 100 (severe pain). Scores converted to 0, 1, 2, or 3 where 0 = no pain and 3 = severe pain.
  Units on a scale | 0.92 (0.85) | 0.71 (0.72) | 0.75 (0.75)
CHAQ - functioning [Mean (Standard Deviation); unit: Units on a scale] — Daily functioning included questions on level of difficulty child had with 8 categories of daily living. Responses ranged from 'without any difficulty' (0) to 'unable to do' (3). Functioning score = sum of highest score in each category divided by number of categories answered; scores ranged from 0 to 3; higher scores indicated more impairment.
  Units on a scale | 0.65 (0.68) | 0.48 (0.54) | 0.52 (0.57)
Number of joints with active arthritis [Mean (Standard Deviation); unit: Joints] — Active arthritis defined as swelling or limitation of motion of the joint accompanied by heat, pain, or tenderness. A total of 36 joints and spine (cervical, thoracic, and lumbar) checked.
  Joints | 3.4 (5.39) | 2.9 (4.14) | 3.0 (4.42)
GISSK - severity of stomach problems [Mean (Standard Deviation); unit: Units on a scale] — GISSK is a validated measure of GI symptom severity and types of GI problems, if any. For severity of stomach problems, participant or caregiver reported severity of participant's stomach problems during the last week using VAS, where scores ranged from 0 (no trouble at all) to 100 (severe stomach problems).
  Units on a scale | 21.9 (25.75) | 12.0 (19.84) | 14.0 (21.47)
Body weight [Median (Full Range); unit: kilogram (kg)] | 33.60 [10.7 to 67.4] | 30.20 [8.7 to 99.5] | 30.90 [8.7 to 99.5]
Height [Median (Full Range); unit: centimeters (cm)] | 141.30 [81.2 to 174.5] | 130.10 [77.5 to 179.0] | 132.00 [77.5 to 179.0]
Body Mass Index (BMI) [Median (Full Range); unit: kilograms per meter squared (kg/m^2)] — Based on World Health Organization (WHO) 2000 Centers for Disease Control growth charts. BMI = Weight in Kilograms divided by (/) (Height in Meters multipled by [*] Height in Meters).
  kilograms per meter squared (kg/m^2) | 17.70 [7.4 to 28.6] | 17.31 [12.5 to 45.1] | 17.55 [7.4 to 45.1]
Weight and Height percentiles overall [Mean (Standard Deviation); unit: Percentile] — Percentile category based on WHO 2000 Centers for Disease Control growth charts
  Percentile
    Weight | 47.22 (29.95) | 56.68 (30.96) | 54.76 (30.94)
    Height | 42.77 (29.59) | 50.70 (30.76) | 49.08 (30.63)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events (AEs) and Serious Adverse Events (SAEs)
Description: Counts of participants who had treatment-emergent adverse events (TEAEs), defined as newly occurring or worsening after first dose. Participants with multiple occurrences of an AE within a category were counted once within the category. AEs attributed to the NSAID (celecoxib or nsNSAID) utilized at time of event, regardless of the initial NSAID treatment at Registry entry.
Time Frame: Baseline up to 2 years
Population: Safety Analysis Set: participants who were prescribed at least one dose of any NSAID. Participants who switched treatment were counted for the NSAID utilized at the time of the event, regardless of the initial NSAID treatment at enrollment.
Measure: Number; unit: Participants
Groups:
- Celecoxib: Participants who received celecoxib at any time during the study. Treatment assignment as per treating physician's judgment. The use and dosage recommendations for celecoxib took place on the basis of the approved Product Label and were adjusted solely according to medical and therapeutic necessity.
- nsNSAIDs: Participants who received nsNSAIDs at any time during the study. Treatment assignment per treating physician's judgment. The use and dosage recommendations for nsNSAIDs took place on the basis of the approved Product Label and were adjusted solely according to medical and therapeutic necessity.
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 68 | 225
Participants
  AEs | 36 | 117
  SAEs | 2 | 9

2. Primary Outcome: JIA Concomitant Medications
Description: JIA medications by class: GI protective agents (eg, proton-pump inhibitors, antacids, surcalfate), other GI, DMARDs, biologics, antihypertensives, NSAIDs (Celecoxib, Diclofenac, Ibuprofen, Meloxicam, Naproxen, other NSAIDs), corticosteroids (oral, IV, intra-articular, other forms), analgesics Acetaminophen, Opioids, other). Participants could receive more than 1 medication.
Time Frame: Year 2 or early termination
Population: Safety Analysis Set subset of participants who received JIA concomitant medications
Measure: Number; unit: Participants
Arm/Group | Celecoxib | nsNSAIDs
Number analyzed (Participants) | 39 | 148
Participants
  GI protective agents | 20 | 54
  Other GI | 5 | 8
  DMARDs | 24 | 102
  Biologics | 13 | 60
  Antihypertensives | 1 | 4
  NSAIDs (Celecoxib) | 7 | 2
  NSAIDs (Diclofenac) | 0 | 0
  NSAIDs (Ibuprofen) | 1 | 9
  NSAIDs (Meloxicam) | 1 | 8
  NSAIDs (Naproxen) | 0 | 7
  NSAIDs (Other) | 0 | 3
  Corticosteroids (oral, IV, intra-articular) | 4 | 15
  Corticosteroids (Other) | 2 | 6
  Analgesics (Acetaminophen, Opioids, Other) | 11 | 19

ADVERSE EVENTS:
Description: Participants who switched treatment were counted for NSAID utilized at time of event, regardless of initial NSAID treatment at enrollment. The same event may appear as both an AE and SAE. However, distinct events are presented.
Groups:
- Celecoxib: Participants who were prescribed celecoxib at any time during the study. Treatment assignment per treating physician's judgment. The use and dosage recommendations for celecoxib took place on the basis of the approved Product Label and were adjusted solely according to medical and therapeutic necessity.
Arm/Group | Celecoxib | nsNSAIDs
Serious Adverse Events (participants affected / at risk) | 2/68 | 9/225
Other Adverse Events (participants affected / at risk) | 35/68 | 114/225
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=68) | nsNSAIDs (N=225)
Febrile Neutropenia (Blood and lymphatic system disorders) | 0 | 1
Agranulocytosis (Blood and lymphatic system disorders) | 0 | 1
Abdominal Pain Lower (Gastrointestinal disorders) | 0 | 1
Condition Aggravated (General disorders) | 1 | 0
Pyrexia (General disorders) | 1 | 0
Cellulitis (Infections and infestations) | 1 | 1
Appendicitis (Infections and infestations) | 0 | 1
Arthritis Bacterial (Infections and infestations) | 0 | 1
Meningitis (Infections and infestations) | 0 | 1
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibrous Histiocytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Migraine (Nervous system disorders) | 1 | 0
Unintended Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Celecoxib (N=68) | nsNSAIDs (N=225)
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 1
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Leukopenia (Blood and lymphatic system disorders) | 0 | 1
Lymphopenia (Blood and lymphatic system disorders) | 0 | 1
Tachycardia (Cardiac disorders) | 1 | 0
Micrognathia (Congenital, familial and genetic disorders) | 1 | 0
Uveitis (Eye disorders) | 0 | 6
Chalazion (Eye disorders) | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 1
Dry eye (Eye disorders) | 0 | 1
Eye Pain (Eye disorders) | 0 | 1
Hypermetropia (Eye disorders) | 0 | 1
Vision Blurred (Eye disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 11 | 28
Abdominal pain (Gastrointestinal disorders) | 9 | 27
Diarrhoea (Gastrointestinal disorders) | 2 | 16
Vomiting (Gastrointestinal disorders) | 5 | 8
Abdominal Pain Upper (Gastrointestinal disorders) | 3 | 9
Constipation (Gastrointestinal disorders) | 2 | 9
Dyspepsia (Gastrointestinal disorders) | 3 | 8
Abdominal Pain Lower (Gastrointestinal disorders) | 1 | 6
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 0 | 6
Stomatitis (Gastrointestinal disorders) | 2 | 4
Mouth Ulceration (Gastrointestinal disorders) | 1 | 2
Abdominal Distension (Gastrointestinal disorders) | 1 | 1
Dry Mouth (Gastrointestinal disorders) | 0 | 2
Faeces Discoloured (Gastrointestinal disorders) | 1 | 1
Faeces Hard (Gastrointestinal disorders) | 0 | 2
Coeliac Disease (Gastrointestinal disorders) | 1 | 0
Crohn's Disease (Gastrointestinal disorders) | 0 | 1
Gastritis (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 0
Disease Progression (General disorders) | 2 | 5
Pyrexia (General disorders) | 0 | 4
Chest Pain (General disorders) | 2 | 0
Drug Intolerance (General disorders) | 0 | 2
Fatigue (General disorders) | 0 | 2
Irritability (General disorders) | 0 | 1
Mucosal Inflammation (General disorders) | 0 | 1
Drug Hypersensitivity (Immune system disorders) | 0 | 1
Hypersensitivity (Immune system disorders) | 0 | 1
Latex Allergy (Immune system disorders) | 0 | 1
Seasonal Allergy (Immune system disorders) | 0 | 1
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 7
Pharyngitis Streptococcal (Infections and infestations) | 1 | 5
Pneumonia (Infections and infestations) | 2 | 2
Sinusitis (Infections and infestations) | 1 | 3
Ear Infection (Infections and infestations) | 1 | 2
Influenza (Infections and infestations) | 2 | 1
Otitis Media (Infections and infestations) | 1 | 2
Pharyngitis (Infections and infestations) | 2 | 1
Viral Infection (Infections and infestations) | 1 | 2
Fungal Skin Infection (Infections and infestations) | 1 | 1
Gastroenteritis (Infections and infestations) | 0 | 2
Tonsillitis (Infections and infestations) | 0 | 2
Adenoiditis (Infections and infestations) | 0 | 1
Bronchitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Chronic Tonsillitis (Infections and infestations) | 1 | 0
Conjunctivitis Infective (Infections and infestations) | 0 | 1
Coxsackie Viral Infection (Infections and infestations) | 0 | 1
Cystitis (Infections and infestations) | 0 | 1
Erythema Infectiosum (Infections and infestations) | 0 | 1
Eye Infection Bacterial (Infections and infestations) | 0 | 1
Eye Infection Viral (Infections and infestations) | 0 | 1
Fungal Infection (Infections and infestations) | 0 | 1
Furuncle (Infections and infestations) | 0 | 1
Gastroenteritis Viral (Infections and infestations) | 0 | 1
Impetigo (Infections and infestations) | 0 | 1
Infection (Infections and infestations) | 1 | 0
Molluscum Contagiosum (Infections and infestations) | 0 | 1
Onychomycosis (Infections and infestations) | 0 | 1
Otitis Externa (Infections and infestations) | 0 | 1
Paronychia (Infections and infestations) | 0 | 1
Rash Pustular (Infections and infestations) | 0 | 1
Staphylococcal Infection (Infections and infestations) | 0 | 1
Streptococcal Infection (Infections and infestations) | 0 | 1
Subcutaneous Abscess (Infections and infestations) | 0 | 1
Tonsillitis Streptococcal (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 6
Arthropod Bite (Injury, poisoning and procedural complications) | 0 | 2
Lower Limb Fracture (Injury, poisoning and procedural complications) | 0 | 1
Weight Decreased (Investigations) | 1 | 1
Blood Pressure Increased (Investigations) | 0 | 1
Blood Urea Increased (Investigations) | 0 | 1
C-reactive Protein Increased (Investigations) | 0 | 1
Hepatic Enzyme Increased (Investigations) | 0 | 1
Red Blood Cell Sedimentation Rate Increased (Investigations) | 0 | 1
Weight Increased (Investigations) | 0 | 1
Anorexia (Metabolism and nutrition disorders) | 3 | 10
Decreased Appetite (Metabolism and nutrition disorders) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 3
Back Pain (Musculoskeletal and connective tissue disorders) | 0 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Growth Retardation (Musculoskeletal and connective tissue disorders) | 0 | 1
Joint Effusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Atrophy (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 | 1
Synovial Cyst (Musculoskeletal and connective tissue disorders) | 0 | 1
Unequal Limb Length (Musculoskeletal and connective tissue disorders) | 1 | 0
Lipoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Headache (Nervous system disorders) | 3 | 9
Dizziness (Nervous system disorders) | 0 | 3
Convulsion (Nervous system disorders) | 0 | 2
Cognitive Disorder (Nervous system disorders) | 0 | 1
Disturbance In Attention (Nervous system disorders) | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Memory Impairment (Nervous system disorders) | 0 | 1
Migraine (Nervous system disorders) | 0 | 1
Paraesthesia (Nervous system disorders) | 0 | 1
Psychomotor Hyperactivity (Nervous system disorders) | 0 | 1
Tremor (Nervous system disorders) | 0 | 1
Attention Deficit/Hyperactivity Disorder (Psychiatric disorders) | 0 | 1
Confusional State (Psychiatric disorders) | 0 | 1
Initial Insomnia (Psychiatric disorders) | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 1
Mood Altered (Psychiatric disorders) | 0 | 1
Sleep Disorder (Psychiatric disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 0 | 3
Urinary Incontinence (Renal and urinary disorders) | 1 | 1
Dysuria (Renal and urinary disorders) | 1 | 0
Proteinuria (Renal and urinary disorders) | 1 | 0
Menstruation Irregular (Reproductive system and breast disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 1 | 0
Vulval Disorder (Reproductive system and breast disorders) | 1 | 0
Asthma Exercise Induced (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea Exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pleuritic Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Postnasal Drip (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Rhinitis Allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 4
Rash (Skin and subcutaneous tissue disorders) | 3 | 2
Eczema (Skin and subcutaneous tissue disorders) | 0 | 3
Pseudoporphyria (Skin and subcutaneous tissue disorders) | 0 | 3
Urticaria (Skin and subcutaneous tissue disorders) | 0 | 2
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 1
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 1
Erythema Multiforme (Skin and subcutaneous tissue disorders) | 0 | 1
Keratosis Pilaris (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Erythematous (Skin and subcutaneous tissue disorders) | 0 | 1
Rash Papular (Skin and subcutaneous tissue disorders) | 1 | 0
Rash Pruritic (Skin and subcutaneous tissue disorders) | 0 | 1
Seborrhoea (Skin and subcutaneous tissue disorders) | 0 | 1
Skin Exfoliation (Skin and subcutaneous tissue disorders) | 0 | 1
Swelling Face (Skin and subcutaneous tissue disorders) | 0 | 1
Vitiligo (Skin and subcutaneous tissue disorders) | 0 | 1
Joint Arthroplasty (Surgical and medical procedures) | 1 | 0
Flushing (Vascular disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Study terminated prematurely: Sponsor released by FDA from post-marketing commitment. As a result, only a small number of participants/analyses could be performed, data must be interpreted with caution. Endpoints arbitrarily assigned as primary.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.